CLINICAL TRIAL: NCT01939990
Title: Nebivolol in Chronic Obstructive Pulmonary Disease
Brief Title: Safety Study of Nebivolol for COPD Patients
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Funding was discontinued.
Sponsor: University of Chicago (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 11-0720
Record Dates: First submitted 2013-01-22; First posted 2013-09-11 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: High Blood Pressure
Keywords: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Hypertension; Pulmonary Disease, Chronic Obstructive | interventions — Nebivolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebivolol (Active Comparator): Group A will be given Nebivolol 5 to 10mg per day
  Interventions: Drug: Nebivolol
- Placebo (Placebo Comparator): Group B will be given Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — The placebo looks like the study drug but it does not contain active ingredients.
  Other Names: Placebo is a sugar pill.
  Arms: Placebo
Drug: Nebivolol — 5 to 10mg per day
  Other Names: bystolic
  Arms: Nebivolol

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of the study drug Nebivolol, in people who suffer with high blood pressure with Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
The study would be a randomized, placebo-controlled trial of 60 hypertensive patients with documented COPD greater than age 40.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of high blood pressure and chronic obstructive pulmonary disease (COPD)

Exclusion Criteria:

* Asthma; Heart failur;
* End stage kidney disease;
* acute myocardial infarction,unstable angina, stroke or TIA within the past year;
* Females who are pregnant, lactating or women of childbearing potential who are not using approved method of contraception.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
to assess blood pressure control | baseline to 4 weeks
  blood pressure control will be assessed per collection of research data at protocol visits.

SECONDARY OUTCOMES:
to assess pulmonary function tests | baseline to 4 weeks
  pulmonary function tests will be assessed at protocol visits

CONTACTS AND LOCATIONS:
Overall Officials: George Bakris, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- See also: clinical trials at the University of Chicago — http://aura.uchicago.edu